CLINICAL TRIAL: NCT06066450
Title: Efficacy of OSFIT Drug-Eluting Stent in Coronary Ostial Artery Stenosis: Multi-center, Prospective, Observational Study (OSFIT Registry)
Brief Title: Efficacy of OSFIT Drug-Eluting Stent in Coronary Ostial Artery Stenosis
Status: Recruiting | Type: Observational
Sponsor: Genoss Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: AJOUIRBOB2023268
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-09

CONDITIONS: Drug-eluting Stent; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OSFITTM drug-eluting stents.: Treatment Group: Group of patients who received treatment with OSFITTM drug-eluting stents.
  Subgroup with OCT (OCT Subgroup): Subgroup of patients who underwent Optical Coherence Tomography (OCT) to verify stent placement accuracy.
  Interventions: Device: Genoss® DES system, Genoss® Osfit system

INTERVENTIONS:
Device: Genoss® DES system, Genoss® Osfit system — This is a drug-eluting stent used to improve the diameter of the coronary artery in patients with symptomatic ischemic heart disease, with de novo lesions in the native coronary artery, where the reference vessel diameter ranges from 2.25mm to 5.00mm.
  Other Names: GENOSS DES(Sirolimus Drug Eluting Coronary Stent) System, Osfit Sirolimus Drug Eluting Coronary Stent System

SUMMARY:
The purpose of this observational study is to evaluate the long-term effectiveness and safety of the OSFIT drug-eluting stent designed to facilitate procedures in coronary artery lesions. Additionally, the study aims to verify the accuracy of stent placement in the lesion of interest using Optical Coherence Tomography (OCT) among subgroups of participants.

The primary endpoint was defined as the composite of target lesion failure (TLF) at the 12-month mark, including cardiac death, target vessel myocardial infarction (MI), or target lesion revascularization.

DETAILED DESCRIPTION:
Investigator plan to enroll a total of 1000 patients who underwent percutaneous coronary intervention (PCI) for coronary artery stenosis within 5mm of the coronary artery ostium using OSFIT drug-eluting stents, with the condition that only GenossTM drug-eluting stents are used if stenting is performed simultaneously in other lesions. These patients will be followed for up to 12 months.

In addition, a subgroup analysis will be conducted using Optical Coherence Tomography (OCT) to assess the accuracy of OSFIT stent placement immediately after the procedure. OCT catheter use will involve the investigation and follow-up of 50 patients each at Ajou University Hospital and Samsung Seoul Hospital. Statistical analysis will involve categorical variables presented as percentages and numbers, compared using the chi-square or Fisher exact test. Continuous variables will be described using means, standard deviations, or medians and interquartile ranges and compared using Student's t-test or the Wilcoxon rank-sum test. The normality of baseline variable distributions will be assessed using histograms, skewness, kurtosis, and the Kolmogorov-Smirnov one-sample test. Kaplan-Meier analysis of cumulative rates of primary and secondary evaluation variables will be performed using the log-rank test.

To identify potential associations with clinical outcomes, all variables showing potential relevance to clinical outcomes will be tested through univariate Cox regression analysis. In order to reduce bias in retrospective studies, a multivariate Cox proportional hazard model will be used to test variables that have a significant impact (p-value < 0.1) in the univariate analysis.

Subgroup analysis will include an imaging analysis of stent insertion adequacy in the group where OCT was performed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 and above.
2. Patients who have voluntarily decided to participate in this study and have provided written consent in accordance with the subject's agreement.
3. Patients who have undergone percutaneous coronary intervention for stenosis within 5mm of the ostium of the coronary artery using OSFITTM drug-eluting stents. (In case of simultaneous stent placement for other lesions, only GenossTM drug-eluting stents should be used.)

Exclusion Criteria:

1. Patients with contraindications to stent treatment and antiplatelet therapy or who have hypersensitivity.
2. Patients with a life expectancy of less than 1 year.
3. Pregnant or lactating women, or those wishing to become pregnant.
4. Patients with ST-elevation myocardial infarction (STEMI).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A patient with stenosis within 5mm of the coronary artery ostium who qualifies for percutaneous coronary intervention with drug-eluting stents
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Targeted lesion failure | 12 months
  A composite of cardiac death, target-vessel MI, or target lesion revascularization

SECONDARY OUTCOMES:
Major adverse cardiovascular events | 12 months
  A composite of all-cause death, MI, or revascularization
All-cause death | 12 months
  All-cause death and cardiac death
Any MI | 12 months
  Any MI and target vessel MI
Any revascularization | 12 months
  Any revascularization and ischemic driven target lesion revascularization
Major bleeding events, BARC 3, 5 | 12 months
  A composite rate of major bleeding events, BARC 3, 5
Any Stroke | 12 months
  Ischemic or hemorrhagic stroke
Any stent thrombosis | 12 months
  efinite or probable stent thrombosis (acute, subacute, late)

CONTACTS AND LOCATIONS:
Overall Officials: seong-jae TaK, MD, PhD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University Hospital, Suwon, South Korea